CLINICAL TRIAL: NCT00281047
Title: The Phase 2 Study of FP-10, the Food Ingredient Derived From Milk Casein, on the Eradication Rates of Helicobacter Pylori by a Triple Therapy With Lansoprazole, Amoxicillin, and Clarithromycin
Brief Title: The Influence of FP-10 on the Eradication Rates of H. Pylori by a Triple Therapy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamamatsu University (Other)
Collaborators: Oita University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hp.FP-10.01
Record Dates: First submitted 2006-01-23; First posted 2006-01-24 (Estimated); Last update posted 2006-01-27 (Estimated); Status verified 2006-01

CONDITIONS: Helicobacter Pylori
Keywords: Helicobacter pylori (H. pylori); FP-10; amoxicillin; clarithromycin; lansoprazole

INTERVENTIONS:
Drug: FP-10

SUMMARY:
FP-10 is a food ingredient derived from milk casein. FP-10 can inhibit H. pylori to attach to the gastric epithelium. FP-10 has been made clear to decrease the intragastric urease activity (which is assumed to be produced by H. pylori) measured by the urea breath test. FP-10 can also detach H. pylori from gastric epithelium. We have hypothesized that FP-10 increases the eradication rates by a triple therapy with a proton pump inhibitor, amoxicillin, and clarithromycin.

DETAILED DESCRIPTION:
H. pylori -positive patients older than 15 years of age with gastritis, gastric ulcer, duodenal ulcer, or gastroduodenal ulcer are invited to participate in the study. These patients had endoscopically and histologically proven ulcers or active chronic gastritis and are all H. pylori-positive. Written informed consent to participation must be obtained from each patient before the study.

During gastroduodenoscopy, biopsy specimens obtained from both the antrum and the corpus of the greater curvature are subjected to the bacterial susceptibility to clarithromycin by culture test or measurements of 23S rRNA mutations at positions 2142 and 2143 (from adenine to guanine).

Patients are treated with 30 mg of lansoprazole bid, 200 mg of clarithromycin bid, and 750 mg of amoxicillin bid for one week. In addition, they take placebo bid, FP10 1 g bid, or FP-10 2 g bid (2 hour after breakfast and at the bed time) for the same one week. Administration of placebo, FP-10 1 g or FP-10 2 g are performed in a double blinded manner.

Eradication of H. pylori was confirmed by a 13C-urea breath test performed one month after eradication therapy. Throughout the study period, the investigators involved in the assessment of H. pylori eradication are blinded to susceptibility to clarithromycin H. pylori strains.

ELIGIBILITY:
Inclusion Criteria:

H. pylori-positive patients who have never undergo the H. pylori eradication therapy -

Exclusion Criteria:

Patients not infected with H. pylori, Patients who are allergic to amoxicillin, clarithromycin, lansoprazole, 13C-urea, or milk casein

-

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 138
Dates: Start 2006-01; Study Completion 2006-05

PRIMARY OUTCOMES:
The effect of FP-01 on the eradication rates of H. pylori infection by a triple therapy

SECONDARY OUTCOMES:
The effect o FP-10 on the eradication rates of clarithromycin-sensitive and -resistant strains of H. pylori by a triple therapy

CONTACTS AND LOCATIONS:
Overall Officials: Takahisa Furuta, MD, PhD, Study Director — Center for Clinical Research, Hamamatsu University School of Medicine; Kazunrai Murakami, MD, PhD, Study Director — Department of Gastroenterology, Oita University Faculty of Medicine; Toshio Fujioka, MD, PhD, Study Chair — Oita University
Locations (7):
- Japan (7):
  - Oita Kouseiren Tsurumi Hospital, Beppu, Oita Prefecture
  - University Hospital of Oita University Faculty of Medicine, Ōita, Oita Prefecture
  - Senoo Clinic for Internal Medicine and Gastroenterology, Hamamatsu, Shizuoka
  - University Hospital of Hamamatsu University School of Medicine, Hamamatsu, Shizuoka
  - Matsushita Clinic, Hamamatsu, Shizuoka
  - Kumagai Clinic for Internal Medicine and Gastroenterology, Hamamatsu, Shizuoka
  - Nakajima Clinic, Kakegawa, Shizuoka

REFERENCES:
- [Background] Furuta T, Sagehashi Y, Shirai N, Sugimoto M, Nakamura A, Kodaira M, Kenmotsu K, Nagano M, Egashira T, Ueda K, Yoneyama M, Ohashi K, Ishizaki T, Hishida A. Influence of CYP2C19 polymorphism and Helicobacter pylori genotype determined from gastric tissue samples on response to triple therapy for H pylori infection. Clin Gastroenterol Hepatol. 2005 Jun;3(6):564-73. doi: 10.1016/s1542-3565(04)00779-7. PMID 15952098
- [Background] Shirai N, Furuta T, Sugimoto M, Nakamura A. [High dose dual PPI/AMPC therapy for the treatment of Helicobacter pylori infection after failure of usual standard triple PPI/AMPC/CAM therapy]. Nihon Rinsho. 2005 Nov;63 Suppl 11:438-41. No abstract available. Japanese. PMID 16363575
- [Background] Okudaira K, Miura S, Furuta T, Sugimoto M, Shirai N. [Concomitant dosing of a H2 receptor antagonist (H2RA) with a triple therapy increases the cure rate of Helicobacter pylori infection]. Nihon Rinsho. 2005 Nov;63 Suppl 11:391-6. No abstract available. Japanese. PMID 16363566
- [Background] Furuta T, Shirai N, Sugimoto M, Nakamura A, Hishida A, Ishizaki T. Influence of CYP2C19 pharmacogenetic polymorphism on proton pump inhibitor-based therapies. Drug Metab Pharmacokinet. 2005 Jun;20(3):153-67. doi: 10.2133/dmpk.20.153. PMID 15988117
- [Background] Furuta T, Shirai N, Sugimoto M, Nakamura A, Okudaira K, Kajimura M, Hishida A. Effect of concomitant dosing of famotidine with lansoprazole on gastric acid secretion in relation to CYP2C19 genotype status. Aliment Pharmacol Ther. 2005 Jul 1;22(1):67-74. doi: 10.1111/j.1365-2036.2005.02523.x. PMID 15963082
- [Background] Okudaira K, Furuta T, Shirai N, Sugimoto M, Miura S. Concomitant dosing of famotidine with a triple therapy increases the cure rates of Helicobacter pylori infections in patients with the homozygous extensive metabolizer genotype of CYP2C19. Aliment Pharmacol Ther. 2005 Feb 15;21(4):491-7. doi: 10.1111/j.1365-2036.2005.02353.x. PMID 15710002
- [Background] Murakami K, Fujioka T. [Drug resistant H. pylori in Japan: general remarks]. Nihon Rinsho. 2005 Nov;63 Suppl 11:198-202. No abstract available. Japanese. PMID 16363531
- [Background] Murakami K, Kodama M, Sato R, Okimoto T, Watanabe K, Fujioka T. Helicobacter pylori eradication and associated changes in the gastric mucosa. Expert Rev Anti Infect Ther. 2005 Oct;3(5):757-64. doi: 10.1586/14787210.3.5.757. PMID 16207167
- [Background] Murakami K, Sato R, Okimoto T, Watanabe K, Nasu M, Fujioka T, Kodama M, Kagawa J. Influence of anti-ulcer drugs used in Japan on the result of (13)C-urea breath test for the diagnosis of Helicobacter pylori infection. J Gastroenterol. 2003;38(10):937-41. doi: 10.1007/s00535-003-1176-x. PMID 14614600
- [Background] Hiramoto S, Itoh K, Shizuuchi S, Kawachi Y, Morishita Y, Nagase M, Suzuki Y, Nobuta Y, Sudou Y, Nakamura O, Kagaya I, Goshima H, Kodama Y, Icatro FC, Koizumi W, Saigenji K, Miura S, Sugiyama T, Kimura N. Melanoidin, a food protein-derived advanced maillard reaction product, suppresses Helicobacter pylori in vitro and in vivo. Helicobacter. 2004 Oct;9(5):429-35. doi: 10.1111/j.1083-4389.2004.00263.x. PMID 15361082
- [Background] Murakami K, Sato R, Okimoto T, Nasu M, Fujioka T, Kodama M, Kagawa J. Efficacy of triple therapy comprising rabeprazole, amoxicillin and metronidazole for second-line Helicobacter pylori eradication in Japan, and the influence of metronidazole resistance. Aliment Pharmacol Ther. 2003 Jan;17(1):119-23. doi: 10.1046/j.1365-2036.2003.01401.x. PMID 12492740
- [Background] Murakami K, Sato R, Okimoto T, Nasu M, Fujioka T, Kodama M, Kagawa J, Sato S, Abe H, Arita T. Eradication rates of clarithromycin-resistant Helicobacter pylori using either rabeprazole or lansoprazole plus amoxicillin and clarithromycin. Aliment Pharmacol Ther. 2002 Nov;16(11):1933-8. doi: 10.1046/j.1365-2036.2002.01368.x. PMID 12390102
- [Background] Murakami K, Nasu M. [Clarithromycin (CAM)]. Nihon Rinsho. 2002 Feb;60 Suppl 2:667-70. No abstract available. Japanese. PMID 11979867
- [Background] Murakami K, Nasu M. [Drug sensitivity test for Helicobacter pylori]. Nihon Rinsho. 2002 Feb;60 Suppl 2:350-3. No abstract available. Japanese. PMID 11979806
- [Background] Murakami K, Fujioka T, Okimoto T, Sato R, Kodama M, Nasu M. Drug combinations with amoxycillin reduce selection of clarithromycin resistance during Helicobacter pylori eradication therapy. Int J Antimicrob Agents. 2002 Jan;19(1):67-70. doi: 10.1016/s0924-8579(01)00456-3. PMID 11814770
- [Background] Asaka M, Satoh K, Sugano K, Sugiyama T, Takahashi S, Fukuda Y, Ota H, Murakami K, Kimura K, Shimoyama T. Guidelines in the management of Helicobacter pylori infection in Japan. Helicobacter. 2001 Sep;6(3):177-86. doi: 10.1046/j.1523-5378.2001.00027.x. PMID 11683920
- [Background] Murakami K, Fujioka T, Kodama R, Kubota T, Tokieda M, Nasu M. Helicobacter pylori infection accelerates human gastric mucosal cell proliferation. J Gastroenterol. 1997 Apr;32(2):184-8. doi: 10.1007/BF02936365. PMID 9085165